CLINICAL TRIAL: NCT06418061
Title: A Multicenter, Open-label, Phase Ia/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IBI3005 in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study of IBI3005 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3005A101
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Unresectable; Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI3005 (Experimental)
  Interventions: Drug: IBI3005

INTERVENTIONS:
Drug: IBI3005 — Bispecific Monoclonal Antibody-Camptothecin Derivative Conjugate for Injection (R & D code: IBI3005)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of IBI3005 and to determine the maximum tolerated dose (MTD) and the recommended Phase 2 Dose (RP2D) of IBI3005.

ELIGIBILITY:
Inclusion Criteria:

Subjects Should have been previously treated with a third-generation EGFR TKI with disease progression. Subjects with positive other driver genes or METex14 mutations are required to undergo targeted therapy and disease progression.

Exclusion Criteria:

Received live vaccines within 4 weeks prior to first administration of the study drug or plan on receiving any live vaccine during the study.Patients are allowed to receive inactivated vaccines.

Uncontrolled diseases including:

* Infection requiring systemic antibiotics, antivirals or antifungals within 2 weeks prior to first dose of the study drug（ antiviral medication for hepatitis B and hepatitis C infection that are compliant with the protocol were allowed）;
* Known human immunodeficiency virus (HIV) infection, or HIV positive (HIV 1/2 Ab positive);
* Acute or chronic active hepatitis B (HbsAg positive and/or HbcAb positive with HBV DNA titer ≥ 104 copies/mL or ≥ 2000 IU/mL or higher than lower limit of detection) or C (HCV Ab positive with HCV RNA titer > 103 copies/mL or higher than lower limit of detection);
* Active COVID-19 infection with obvious symptoms requiring treatment or hospitalization, such as pyrexia, dyspnea, nausea, vomiting, diarrhea, etc.;
* Active tuberculosis infection, or still on anti-tuberculosis therapy or received anti tuberculosis therapy within 1 year prior to first administration of the study drug;
* Active syphilis infection or latent syphilis requiring treatment;
* Symptomatic congestive heart failure Grade II-IV (New York Heart Association [NYHA]), symptomatic or uncontrolled arrhythmias, QTc interval > 480 ms or personal or family history of congenital long/short QT syndrome;
* Hypertension that does not receive standardized therapy or still uncontrollable hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg); Any history of life-threatening hemorrhage, or hemorrhage requiring (including but not limited to gastrointestinal bleeding, hemoptysis, etc) blood transfusion, endoscopy, or surgery, within 3 months prior to the first administration of study drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of subjects with adverse events | Up to 3 years
  defined as any untoward medical occurrence, whether or not there is a causal relationship with the study drug, in a clinical study subject from the time informed consent form is signed
Number of subjects with clinically significant changes in physical examination results | Up to 3 years
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in vital signs | Up to 3 years
  Vital signs including body temperature, pulse, respiratory rate, SpO2 and blood pressure
Dose limiting toxicities (DLTs) | Up to 4 weeks
  Dose limiting toxicities (DLTs) to establish MTD and/or RP2D.

SECONDARY OUTCOMES:
area under the curve (AUC) | up to 3 years
  area under the curve (AUC) of single and multiple doses of IBI3005
maximum concentration (Cmax) | up to 3 years
  maximum concentration (Cmax) of single and multiple doses of IBI3005
time to maximum concentration (Tmax) | up to 3 years
  time to maximum concentration (Tmax) of single and multiple doses of IBI3005
clearance (CL) | up to 3 years
  clearance (CL) of single and multiple doses of IBI3005
apparent volume of distribution (V) | up to 3 years
  apparent volume of distribution (V) of single and multiple doses of IBI3005
half-life (t1/2) | up to 3 years
  half-life (t1/2) of IBI3005 to the last administration of IBI3005
anti-drug antibody (ADA) | up to 3 years
  Incidence and characterization of anti-drug antibody (ADA).
objective response rate (ORR) | up to 3 years
  objective response rate (ORR) as evaluated per the RECIST v1.1 criteria.
duration of response (DoR) | up to 3 years
  duration of response (DoR) as evaluated per the RECIST v1.1 criteria.
time to response (TTR) | up to 3 years
  time to response (TTR) as evaluated per the RECIST v1.1 criteria.
progression free survival (PFS) | up to 3 years
  as evaluated per the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital & Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No